CLINICAL TRIAL: NCT07006337
Title: Surgical Operating Room Enhancement Curriculum for Medical Students: A Quality Improvement and Prospective Cohort Study
Brief Title: Surgical Operating Room Enhancement Curriculum for Medical Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Richard Hsu, Resident Physician, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-24-06-6938
Record Dates: First submitted 2025-05-15; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Gynecology; Medical Education; Operating Rooms

STUDY DESIGN:
Intervention Model Description: The study uses a prospective, parallel-group design. Medical students are stratified by their clinical rotation cohorts (5-week blocks) to ensure baseline equivalence in knowledge and experience. Each cohort is assigned either to the intervention or control arm for the duration of their rotation. The intervention group participates in the enrichment course, while the control group completes the standard rotation. Both groups complete knowledge and perception assessments at the end of their respective rotations
Masking Description: Not applicable. Participants, care providers, and investigators will be aware of group assignments due to the nature of the educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Operating Room Enrichment Course (Experimental): Participants in this arm will receive the enhanced Surgical Operating Room (OR) Enrichment Course as part of their medical student curriculum. This intervention includes both didactic lectures led by gynecology-trained physicians. The curriculum covers preoperative evaluation, perioperative complication prevention, gynecologic anatomy, surgical techniques, gynecologic emergencies, operative decision-making, postoperative care, and OR tasks and procedures. Participants will complete pre- and post-intervention surveys to assess changes in knowledge, proficiency, and clinical perceptions related to gynecologic surger
  Interventions: Other: Surgical Operating Room Enrichment Course
- Standard Curriculum (Control) (Active Comparator): Participants in this arm will follow the standard medical student curriculum for the gynecology rotation, without the additional enrichment course. At the end of their rotation, they will complete a questionnaire assessing their baseline knowledge and perceptions of gynecologic surgery. No additional didactic or hands-on surgical skills training beyond the standard curriculum will be provided to this group
  Interventions: Other: Active Comparator #1

INTERVENTIONS:
Other: Surgical Operating Room Enrichment Course — The intervention consists of multiple structured training sessions delivered during the gynecology rotation. Sessions include lectures on surgical principles and gynecologic procedures. The course is taught by OBGYN physicians and is designed to enhance students' proficiency in surgical techniques, perioperative care, and management of gynecologic emergencies. Educational materials are based on relevant surgical guidelines and textbooks
  Arms: Surgical Operating Room Enrichment Course
Other: Active Comparator #1 — Active Comparator #1
  Arms: Standard Curriculum (Control)

SUMMARY:
The goal of this clinical trial is to assess whether integrating an enhanced Surgical Operating Room (OR) curriculum into the medical student program improves knowledge and proficiency in gynecologic surgical techniques and procedures among medical students at Wayne State University. The main questions it aims to answer are:

Does the Surgical Operating Room Enrichment Course increase medical students' knowledge and comfort with gynecologic surgical procedures?

Does participation in the course improve students' clinical perceptions and management of gynecologic emergencies?

Researchers will compare students who participate in the Surgical Operating Room Enrichment Course (intervention group) to those who complete the standard rotation (control group) to see if the enhanced curriculum leads to greater improvements in knowledge and clinical skills.

Participants will:

Attend virtual didactic lectures covering gynecologic anatomy, perioperative care, surgical techniques, and management of gynecologic emergencies

Complete pre- and post-training surveys assessing knowledge, skills, and perceptions related to gynecologic surgery

This study involves approximately 60 medical students, with participation being voluntary and all responses de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Medical students currently enrolled in the Wayne State University OBGYN clinical rotation (5-week block)
* Willingness to voluntarily participate in surveys and training sessions
* Ability to attend all didactic lectures

Exclusion Criteria:

* Prior completion of a structured surgical operating room enrichment course (e.g., elective subspecialty training)
* Inability to participate virtual sessions due to conflicting clinical/academic schedules
* Non-English speakers (due to English-language survey instruments)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge and Proficiency in Gynecologic Surgical Techniques | From baseline (start of rotation) to end of rotation (5 weeks)
  Assessed by the difference in scores on a validated knowledge and skills questionnaire administered before and after participation in the Surgical Operating Room Enrichment Course. The questionnaire evaluates understanding of gynecologic anatomy, surgical steps, perioperative care, and technical proficiency, using a combination of multiple-choice, Likert scale, and open-ended questions. Improvement will be measured by comparing pre- and post-intervention scores within and between the intervention and control groups.

SECONDARY OUTCOMES:
Change in Clinical Perceptions and Comfort with Gynecologic Emergencies | From baseline (start of rotation) to end of rotation (5 weeks)
  Measured by the difference in self-reported confidence and comfort levels in managing gynecologic emergencies, as captured by Likert scale items and open-ended responses in the pre- and post-intervention surveys. This outcome will assess whether the enrichment course influences students' perceived preparedness for real-world clinical scenarios.
Participant Satisfaction with Surgical Operating Room Curriculum | At end of rotation (5 weeks)
  Assessed via post-intervention survey items evaluating satisfaction with the curriculum content, teaching methods, and perceived educational value. Survey includes Likert scale and open-ended feedback questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University SOM, Dept of OBGYN, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data,including data dictionaries, survey responses, and outcome measures, will be shared with qualified researchers for independent scientific research, following publication of the main results. No personal identifiers or protected health information (PHI) will be included.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the main results and for up to 36 months thereafter.
Access Criteria: Access to IPD and supporting documents will be granted to qualified researchers with an approved research proposal and statistical analysis plan. Requestors must sign a data sharing agreement too. Requests can be submitted to the principal investigator via institutional contact.